CLINICAL TRIAL: NCT06669364
Title: Retrospective Analysis of Routine EEG to Validate a Computational Biomarker (BioEP) as an Assessment Aid for Seizure Susceptibility.
Brief Title: A Retrospective Study to Validate BioEP as an Assessment Aid for Seizure Susceptibility
Acronym: SOLITAIRE
Status: Not yet recruiting | Type: Observational
Sponsor: Neuronostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NNBioEP003
Record Dates: First submitted 2024-08-07; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epilepsy: Device: BioEP
  All patient's EEG will have the BioEP score conducted on it
- Non-epilepsy: Device: BioEP
  All patient's EEG will have the BioEP score conducted on it

SUMMARY:
The goal of this retrospective study is to validate BioEP during routine adult EEG recording in an outpatient setting, using patients with a known epilepsy diagnosis. The main objectives of the study are:

* To validate BioEP during routine adult EEG recording in an outpatient setting, using patients with a known diagnosis
* To examine whether the use of BioEP could support a more efficient patient pathway to diagnosis (thus adding economic value), by reducing time to final diagnosis and/or the number of clinical appointments needed.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 22 and above) who had a routine EEG in an outpatient setting, following a suspected seizure.
* A diagnosis of epilepsy or alternate condition has been reached. A period of at least 3 years has passed since ultimate diagnosis, which itself has remained stable.
* EEGs performed to ABRET & IFCN standards using a minimum of 19 electrodes and additional technical requirements.

Exclusion Criteria:

* Subject was not suspected of having had a seizure or epilepsy.
* Subject has a dual diagnosis of epilepsy AND non-epileptic seizures.
* Subject's final diagnosis unknown, unstable, or less than three years passed since an unchanged diagnosis was made.
* Incomplete or unreliable metadata, such as the age, sex, and treatment status at the time of the EEG recording.
* Sleep deprived EEG recordings in the outpatient setting.
* Encephalopathic subjects.
* Poor quality EEGs (multiple artefacts) that do not fulfil technical criteria for analysis.
* Known structural abnormalities or skull breaches, including historical cases, or with people with metal or plastic implants in their brain or skull.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population with a diagnosis of epilepsy
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
To validate BioEP during routine adult EEG recording in an outpatient setting, using patients with a known diagnosis | 6 months
  Diagnostic accuracy, defined by a primary endpoint family1 of two ranked endpoints. Specifically, we are testing whether BioEP has superior sensitivity to initial EEG alone and is no worse than EEG alone for specificity (non-inferiority). These are ranked hypotheses with sensitivity taking precedence (fixed sequence method) . That is, we shall only proceed to comparing specificity if sensitivity is superior.

SECONDARY OUTCOMES:
To examine whether the use of BioEP could support a more efficient patient pathway to diagnosis | 6 months
  To assess if BioEP can positively influence the patient pathway by reducing number of clinical appointments to diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Milaana Mainstone, Study Director — Neuronostics Ltd